CLINICAL TRIAL: NCT05406583
Title: A Phase I Study of the Safety, Tolerability, and Pharmacokinetics of Dolutegravir in Neonates Exposed to HIV-1
Brief Title: A Study of the Safety, Tolerability, and Pharmacokinetics of Dolutegravir in Neonates Exposed to HIV-1
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: ViiV Healthcare (Industry); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: IMPAACT 2023; 38637 (Other: DAIDS Study ID)
Record Dates: First submitted 2022-06-01; First posted 2022-06-06 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-07

CONDITIONS: HIV
Keywords: Antiretroviral; Dolutegravir; Newborn; Infant; HIV/AIDS; Perinatal; Pharmacokinetics; Prophylaxis; Prevention; Safety
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — dolutegravir; Suspensions

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort 1 (Experimental): Cohort 1 will be opened first to accrual, with Strata 1A and 1B being opened concurrently, to evaluate the PK and safety of two single DTG liquid suspension doses for the relevant stratum. Stratum 1C will only be opened to accrual if PK and safety data from Strata 1A and 1B infants support administration of DTG 5 mg DT across all neonates, or only in neonates with a minimum birth weight.
  * Stratum 1A (DTG-naïve): Infants with no in utero exposure to maternal DTG (no exposure to DTG during the two weeks prior to delivery)
  * Stratum 1B (DTG-exposed): Infants with in utero exposure to maternal DTG (mothers who receive at least one dose of DTG within 72 hours prior to delivery)
  * Stratum 1C (DTG-naïve): Infants with no in utero exposure to maternal DTG (no exposure to DTG during the two weeks prior to delivery).
  Interventions: Drug: Dolutegravir 0.5 mg/kg oral suspension; Drug: Dolutegravir 5 mg Dispersible Tablets
- Cohort 2 (Experimental): Cohort 2, Strata 2A and 2B, will be opened to accrual when the DTG dose and formulation to be administered for each stratum are established based on the PK and safety data from all Cohort 1 strata (Strata 1A and 1B, and 1C if applicable) and available data from other studies.
  * Stratum 2A (DTG-naïve): Infants with no in utero exposure to maternal DTG (no exposure to DTG during the two weeks prior to delivery)
  * Stratum 2B (DTG-exposed): Infants with in utero exposure to maternal DTG (mothers who receive at least one dose of DTG within 72 hours prior to delivery)
  Interventions: Drug: Dolutegravir 0.5 mg/kg oral suspension; Drug: Dolutegravir 5 mg Dispersible Tablets

INTERVENTIONS:
Drug: Dolutegravir 0.5 mg/kg oral suspension — DTG 0.5 mg/kg liquid suspension administered orally
  Other Names: DTG
Drug: Dolutegravir 5 mg Dispersible Tablets — DTG 5 mg DT administered orally

SUMMARY:
This study will test an anti-HIV drug (ARV) for newborn babies. The study will include a minimum of 36 and up to 108 mothers living with HIV and their newborn babies from Brazil, South Africa, Thailand, and the United States. Infants will be in the study for approximately 16 weeks (four months) after they are born. Mothers will not receive study drug and will exit the study after the Entry visit.

ELIGIBILITY:
Inclusion Criteria:

1. Mother is of legal age or circumstance to provide independent informed consent and is willing and able to provide written informed consent for her and permission for her infant's participation in this study.
2. Mother has confirmed HIV-1 infection based on positive test results from two samples collected from two separate blood collection tubes per Sample #1 and Sample #2 protocol requirements. Test results may be obtained from medical records or from testing performed during the study screening period:

   * For results obtained from medical records, adequate source documentation, including the date of specimen collection, date of testing or date of test result, name of test/assay performed, and test result, must be available in study records prior to study entry. Requirements related to laboratory operations (e.g., CLIA, GCLP, or VQA) and related to regulatory authority (e.g., FDA) approvals do not apply to results obtained from medical records.
   * If adequate source documentation is not available, Sample #1 and/or Sample #2 should be collected during the study screening period and tested in the site's designated testing laboratory. If both samples are tested using antibody tests, at least one of the samples must be tested in a laboratory that operates according to CLIA or equivalent (for US sites) or GCLP (for non-US sites) guidelines and participates in an appropriate external quality assurance program. If nucleic acid testing is used, at least one test must be performed in the site's CLIA-certified or equivalent (for US sites) or VQA-certified (for non-US sites) laboratory.
   * All study-specific samples tested to determine HIV-1 status must be whole blood, serum, or plasma. HIV testing methods and algorithms must be approved for each site by the IMPAACT Laboratory Center (for NIAID-funded sites) or Westat (for NICHD-funded sites). All test methods should be FDA-approved, if available.
3. At entry, infant meets DTG exposure requirements, based on mother's report and confirmed by medical records if available, as follows:

   * For Cohort 1, Strata 1A and 1C, and Cohort 2, Stratum 2A: Infant born to a mother who did not receive DTG during the two weeks immediately prior to delivery.
   * For Cohort 1, Stratum 1B, and Cohort 2, Stratum 2B: Infant born to a mother who received at least one dose of DTG less than or equal to 72 hours prior to delivery.
4. Infant was singleton with a gestational age at birth of at least 37 weeks.
5. At birth, infant's weight was as follows:

   * For Cohort 1, Strata 1A and 1B, and Cohort 2, Strata 2A and 2B: At least 2 kg
   * For Cohort 1, Stratum 1C:

     1. At least 2 kg
     2. At least 3 kg
6. At screening, infant has the following laboratory test results

   * ALT (normal)
   * AST (normal or Grade 1)
   * Total bilirubin (normal or Grade 1)
   * Hemoglobin (normal, Grade 1, or Grade 2)
   * White blood cells (normal, Grade 1, or Grade 2)
   * Platelets (normal, Grade 1, or Grade 2)
   * Creatinine (normal, Grade 1, or Grade 2)
7. At entry, infant is less than or equal to five days of life.
8. At entry, infant has initiated standard of care ARV prophylaxis (i.e., received at least one dose of ARV regimen prior to entry).
9. At entry, infant is generally healthy as determined by the site investigator based on review of all available medical history information and physical examination findings.

Exclusion Criteria:

1. Known maternal-fetal blood group incompatibility as evidenced by the presence of an unexpected clinically significant maternal red blood cell antibody that is known to cause hemolytic disease of the fetus and newborn.
2. Infant or breastfeeding mother is receiving any disallowed medication.
3. At entry, infant with a documented positive HIV nucleic acid test result.
4. Infants with prior exchange transfusion or with elevated bilirubin that would require exchange transfusion.
5. Mother or infant has any condition that, in the opinion of the site investigator or designee, would make participation in the study unsafe, complicate interpretation of study outcome data, or otherwise interfere with achieving the study objectives.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2022-10-05 (Actual); Primary Completion 2025-03-12 (Actual); Study Completion 2025-05-22 (Actual)

PRIMARY OUTCOMES:
Proportion of infants classified as "study drug-related" safety failures. | Initial study drug dosing through 2 weeks after off treatment date
  An infant is classified as a "study drug-related" safety failure for the primary safety study objective if any of the following occurred after the initial study drug dosing through two weeks after permanent discontinuation of the study drug (i.e., two weeks after off treatment date):
  * Grade 3 or 4 AE assessed as related to study drug, or
  * Death (Grade 5 AE) assessed as related to the study drug, or
  * Life-threatening AE assessed as related to study drug, or
  * AE assessed as related to study drug that leads to premature permanent discontinuation of the study drug.
Proportion of infants classified as safety failures. | Initial study drug dosing through 2 weeks after off treatment date
  An infant is classified as a safety failure for the primary safety study objective if any of the following occurred after the initial study drug dosing through two weeks after permanent discontinuation of the study drug (i.e., two weeks after off treatment date):
  * Grade 3 or 4 AE, or
  * Death (Grade 5 AE)
Proportion of infants who are not able to tolerate the study drug. | Initial study drug dosing through study drug discontinuation
  An infant is considered not able to tolerate the study drug if the infant experiences problems taking the study drug or experiences any AE assessed as related to study drug that leads to premature permanent discontinuation of the study drug.
C(last) for DTG | 28 months
Area under the curve (AUC) for DTG | 28 months
C(trough) for DTG | 28 months
AUC(0-tau) for DTG | 28 months

SECONDARY OUTCOMES:
Proportion of infants classified as "study drug-related" safety failures. | Initial study drug dosing through Week 16
  An infant is classified as a "study drug-related" safety failure for the secondary study safety objective if any of the following occurred after the initial study drug dosing through Week 16:
  * Grade 3 or 4 AE assessed as related to study drug, or
  * Death (Grade 5 AE) assessed as related to the study drug, or
  * Life-threatening AE assessed as related to study drug, or
  * AE assessed as related to study drug that leads to premature permanent discontinuation of the study drug.
Proportion of infants classified as safety failures. | Initial study drug dosing through Week 16
  An infant is classified as a safety failure for the secondary study safety objective if any of the following occurred after the initial study drug dosing through Week 16:
  * Grade 3 or 4 AE, or
  * Death (Grade 5 AE)

OTHER OUTCOMES:
Association of UGT1A1 gene sequence variants with DTG CL/F | 28 months

CONTACTS AND LOCATIONS:
Overall Officials: Diana Clarke, Pharm.D., Study Chair — BMC/Dept. of Pharmacy
Locations (15):
- United States (8):
  - USC - Maternal Child Adolescent/Adult Center, Los Angeles, California
  - David Geffen School of Medicine at UCLA NICHD CRS, Los Angeles, California
  - University of Colorado Denver NICHD CRS, Aurora, Colorado
  - Emory University School of Medicine NICHD CRS, Atlanta, Georgia
  - Rush University, Cook County Hospital NICHD CRS, Chicago, Illinois
  - Bronx-Lebanon Hospital Center NICHD CRS, The Bronx, New York
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - Baylor College of Medicine/ Texas Children's Hospital NICHD CRS, Houston, Texas
- South Africa (4):
  - Soweto, Johannesburg, Gauteng
  - Wits RHI Shandukani Research Centre CRS, Johannesburg, Gauteng
  - Umlazi, Durban, KwaZulu-Natal
  - FAMCRU, Cape Town
- Thailand (3):
  - Siriraj Hospital, Mahidol University NICHD CRS, Bangkok
  - Chiang Mai University HIV Treatment, Chiang Mai
  - Chiangrai Prachanukroh Hospital NICHD CRS, Chiang Rai

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie results in the publication, after deidentification.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 3 months following publication and available throughout period of funding of the International Maternal Pediatric Adolescent AIDS Clinical Trial (IMPAACT) Network by NIH.
Access Criteria: * With whom? Researchers who provide a methodologically sound proposal for use of the data that is approved by the IMPAACT Network.
  * For what types of analyses? To achieve aims in the proposal approved by the IMPAACT Network.
  * By what mechanism will data be made available? Researchers may submit a request for access to data using the IMPAACT "Data Request" form at: https://www.impaactnetwork.org/resources/study-proposals.htm. Researchers of approved proposals will need to sign an IMPAACT Data Use Agreement before receiving the data.
URL: http://www.impaactnetwork.org/